CLINICAL TRIAL: NCT03349567
Title: The Use of Audit-and-Feedback to Improve Antimicrobial-Prescribing in Emergency Departments: a Quasi-experimental Study
Brief Title: Improving Antimicrobial-Prescribing in Emergency Departments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa City Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Daniel Livorsi, Physician-investigator, Iowa City Veterans Affairs Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 201708772
Record Dates: First submitted 2017-11-17; First posted 2017-11-21 (Actual); Results first posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Anti-Bacterial Agents; Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Audit-and-feedback (Experimental): The experimental arm will consist of Emergency Department providers who do receive the intervention.
  Interventions: Behavioral: Audit-and-feedback
- Control (No Intervention): The control arm will consist of providers who do not receive the intervention.

INTERVENTIONS:
Behavioral: Audit-and-feedback — We will monitor the antimicrobial-prescribing of providers in the experimental arm. Our study team will meet with providers in the experimental arm to provide guidance on optimal antimicrobial-prescribing. We will provide personalized feedback to providers in the experimental arm once every quarter.
  Other Names: Academic detailing
  Arms: Audit-and-feedback

SUMMARY:
Antimicrobial resistance is one of today's most urgent public health problems. One of the most important strategies to slow the spread of antimicrobial resistance is the promotion of judicious antimicrobial use. There are tremendous opportunities to reduce unnecessary antimicrobial-prescribing, particularly in Emergency Departments (EDs). In this study, the investigators will work collaboratively with ED providers in the Veterans Health Administration (VHA) to reduce unnecessary antimicrobial use. Academic-detailing and an audit-and-feedback intervention will be implemented, and the study will assess how overall antimicrobial-prescribing changes once these interventions are performed. ED providers will be shown how their antimicrobial-prescribing compares to their peers, thereby encouraging them to consider their professional reputation when making prescribing decisions. To assess the impact of this intervention, the study will monitor providers' antimicrobial-prescribing behavior through an automated metric, i.e. number of antimicrobial prescriptions per number of patient-visits. To assess changes in the appropriateness of antimicrobial-prescribing, the study team will also perform manual chart reviews and compare prescribing decisions to published guidelines.

DETAILED DESCRIPTION:
Using a quasi-experimental design, the study team will work collaboratively with ED providers in the Veterans Health Administration (VHA) to improve antimicrobial-prescribing. Academic-detailing and an audit-and-feedback intervention will be implemented. Through audit-and-feedback, providers will be shown how their antimicrobial-prescribing compares to their peers, thereby encouraging them to consider their professional reputation when making prescribing decisions.

The study will use a pretest-posttest design (quasi-experimental design with a non-equivalent control group) to assess the effect of our pilot intervention at 2 participating EDs and 2 control EDs. For each ED, the pretest period will be the 12 months prior to the intervention. The intervention itself will last 12 months.

There will be an estimated 30 ED providers at the 2 study sites and 30 ED providers at the 2 control sites. Only antimicrobial prescriptions to patients discharged from the ED will be evaluated.

The primary outcome will be antimicrobial-prescribing volume adjusted for the total number of patient-visits. Secondary outcomes include the frequency of guideline-discordant antimicrobial-prescribing and adverse events.

At the conclusion of the pilot trial, a quasi-experimental interrupted time-series (ITS) analysis will be performed to assess the change in monthly antimicrobial usage for the 2 intervention sites combined and the 2 control sites combined. The time frame for this ITS analysis will be the one-year prior to the pilot trial's initiation through the trial's 1-year intervention period for a total of 24 months. In addition, a multivariable analysis will be performed to identify predictors of guideline-discordant therapy.

ELIGIBILITY:
Inclusion Criteria:

--An ED provider at one of the intervention or control sites.

Exclusion Criteria:

--An ED provider who sees less than 100 patients in the ED per year.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Richard Roudebush VAMC, Indianapolis, Indiana
  - Sioux Falls VA, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We performed a quasi-experimental study with an interrupted time-series design and a matched-pair non-equivalent control group. There were 2 intervention sites and 2 control sites; 27/31 providers were enrolled at intervention sites. We measured outcomes in the PATIENTS seen at these 4 EDs. In a difference-in-differences analysis, outcomes were compared across intervention and control sites in patients seen before the intervention period (i.e. baseline) to those during the intervention period.
Groups:
- Audit-and-feedback: The experimental arm will consist of 2 Emergency Departments. We will attempt to enroll all ED providers at our 2 intervention sites, and for the analysis, site-level data will be used.
  Audit-and-feedback: We will monitor the antimicrobial-prescribing of providers in the experimental arm. Our study team will meet with providers in the experimental arm to provide guidance on optimal antimicrobial-prescribing. We will provide personalized feedback to providers in the experimental arm once every quarter.
- Control: The control arm will consist of 2 ED sites that do not receive the intervention. For the analysis, the control sites will be analyzed at the site-level.
Period: Overall Study
Arm/Group | Audit-and-feedback | Control
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: These numbers reflect patients seen in the 4 participating EDs during the baseline and intervention periods.
Groups:
- Patients Seen in the ED at Audit-and-feedback Sites During the Intervention Period: These measures reflect patients seen at audit-and-feedback sites during the intervention period.
- Patients Seen in the ED at Control Sites During the Intervention Period: These baseline measures reflect patients seen at control sites during the intervention period.
- Patients Seen in the ED at Audit-and-feedback Sites During the Baseline Period: These measures reflect patients seen at audit-and-feedback sites before the intervention period, i.e. during the baseline period.
- Patients Seen in the ED at Control Sites During the Baseline Period: These measures reflect patients seen at control sites before the intervention period, i.e. during the baseline period.
- Total: Total of all reporting groups
Arm/Group | Patients Seen in the ED at Audit-and-feedback Sites During the Intervention Period | Patients Seen in the ED at Control Sites During the Intervention Period | Patients Seen in the ED at Audit-and-feedback Sites During the Baseline Period | Patients Seen in the ED at Control Sites During the Baseline Period | Total
Number analyzed (Participants) | 23164 | 28835 | 28016 | 33077 | 113092
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [59 to 62] | 60 [59 to 61] | 60 [58 to 62] | 60 [59 to 60] | 60 [59 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2532 | 2627 | 3014 | 3159 | 11332
  Male | 20,632 | 26208 | 25002 | 29918 | 101760
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 204 | 336 | 243 | 361 | 1144
  Asian | 39 | 190 | 70 | 218 | 517
  Native Hawaiian or Other Pacific Islander | 55 | 125 | 94 | 158 | 432
  Black or African American | 5106 | 2720 | 5990 | 3215 | 17031
  White | 16343 | 23832 | 19893 | 27323 | 87391
  More than one race | 321 | 403 | 389 | 467 | 1580
  Unknown or Not Reported | 1096 | 1229 | 1337 | 1335 | 4997
% of total visits prescribed an antimicrobial (monthly median) [Median (Inter-Quartile Range); unit: Percentage of visits prescribed an abx] | 19.1 [17.8 to 20.4] | 21.6 [19.9 to 22.4] | 21.2 [20.3 to 23.7] | 20.9 [19.4 to 23.4] | 20.7 [19.4 to 22.5]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patient-visits Prescribed an Antimicrobial at Their ED Visit
Description: This outcomes is defined as the total number of antimicrobial-prescribing visits divided by the total number of patient-visits. This metric will be calculated on a monthly basis for each site (2 intervention, 2 control). It will be calculated during the baseline and intervention periods. Therefore, each site will contribute 24 data points.
Time Frame: This outcome will be calculated every month during the baseline and intervention periods. An interrupted time-series analysis will be performed to evaluate how this monthly percentage changed after the intervention period began.
Population: For the Outcome Measure Data Table shown below, patient-visits were stratified by period (i.e. baseline and intervention period), and outcomes were compared across these two periods between intervention and control sites. Please see our statistical analysis plan for further details. For the intervention and control sites, the "overall number of participants analyzed" in the Arms/Groups table equals the sum of the "number analyzed" for the baseline and intervention periods, as shown below.
Measure: Number; unit: percentage of visits prescribed an abx
Groups:
- Patients Seen in the ED at Audit-and-feedback Sites: All patients seen in the ED at audit-and-feedback sites will be considered to have been exposed during the intervention.
- Patients Seen in the ED at Control Sites: All patients seen in the ED at audit-and-feedback sites will be considered to not have been exposed to the intervention.
Arm/Group | Patients Seen in the ED at Audit-and-feedback Sites | Patients Seen in the ED at Control Sites
Number analyzed (Participants) | 51180 | 61,912
percentage of visits prescribed an abx
  Baseline: number analyzed (Participants) | 28016 | 33077
  Baseline | 21.2 | 20.9
  Intervention period: number analyzed (Participants) | 23164 | 28835
  Intervention period | 19.1 | 21.6
Statistical Analysis 1: Comparison: Patients Seen in the ED at Audit-and-feedback Sites vs Patients Seen in the ED at Control Sites; Test type: Superiority; p = 0.35, Mixed Models Analysis; Segmented regression analysis was conducted using generalized linear models to estimate change in monthly antimicrobial prescription rates; Incident rate ratio = 0.99, 95% CI 2-sided [0.98 to 1.01]

2. Secondary Outcome: Percentage of Patient-visits Prescribed a Late Antimicrobial Prescription More Than 24 Hours After But Within 30 Days of Their ED Visit
Description: Late antimicrobial prescription is defined as the prescription of an (additional) antimicrobial by any provider more than 24 hours after but within 30 days of the patient's ED visit.
Time Frame: For both intervention and control sites, the outcome will be reported as a monthly median, which is calculated across the 12 baseline and the 12 intervention months.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of visits exposed to late abx
Arm/Group | Patients Seen in the ED at Audit-and-feedback Sites | Patients Seen in the ED at Control Sites
Number analyzed (Participants) | 51180 | 61912
percentage of visits exposed to late abx
  Baseline: number analyzed (Participants) | 28016 | 33077
  Baseline | 31.5 [28.6 to 36.1] | 29.5 [26.5 to 31.9]
  Intervention: number analyzed (Participants) | 23164 | 28835
  Intervention | 31.1 [28.6 to 35.8] | 28.5 [25.4 to 32.5]
Statistical Analysis 1: Comparison: Patients Seen in the ED at Audit-and-feedback Sites vs Patients Seen in the ED at Control Sites; Test type: Non-Inferiority — A Poisson regression model with log link was used to estimate the rate of safety outcomes. Models were adjusted for time as a continuous covariate, an indicator for month of implementation of intervention (Oct 2018), and included random effects to account for repeated measurements. An interaction variable for the study period (baseline or intervention) and site (intervention or control) was included in the model to estimate the Incident Rate Ratio (IRR) and 95% CIs; Incident rate ratio = 1.12, 95% CI 2-sided [0.93 to 1.35]

3. Secondary Outcome: Percentage of Patient-visits Who Were Hospitalized More Than 24 Hours After But Within 30 Days of Their ED Visit
Description: Hospitalization is defined as the need for hospitalization for any indication at a VA-facility more than 24 hours after but within 30 days of the patient's index visit to the ED.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of visits hospitalized
Arm/Group | Patients Seen in the ED at Audit-and-feedback Sites | Patients Seen in the ED at Control Sites
Number analyzed (Participants) | 51180 | 61912
percentage of visits hospitalized
  Baseline: number analyzed (Participants) | 28016 | 33077
  Baseline | 5.9 [4.9 to 6.5] | 5.6 [4.9 to 6.1]
  Intervention period: number analyzed (Participants) | 23164 | 28835
  Intervention period | 5.9 [5.1 to 6.6] | 5.8 [5.2 to 6.3]
Statistical Analysis 1: Comparison: Patients Seen in the ED at Audit-and-feedback Sites vs Patients Seen in the ED at Control Sites; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Incident rate ratio = 1.01, 95% CI 2-sided [0.81 to 1.27]

4. Secondary Outcome: Percentage of Patient-visits Who Died More Than 24 Hours After But Within 30 Days of Their ED Visit
Description: Death is defined as all-cause death more than 24 hours after and within 30-days of the patient's ED visit.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of patient-visits who died
Arm/Group | Patients Seen in the ED at Audit-and-feedback Sites | Patients Seen in the ED at Control Sites
Number analyzed (Participants) | 51180 | 61912
percentage of patient-visits who died
  Baseline: number analyzed (Participants) | 28016 | 33077
  Baseline | 0.56 [0.4 to 0.7] | 0.61 [0.4 to 0.8]
  Intervention period: number analyzed (Participants) | 23164 | 28835
  Intervention period | 0.60 [0.4 to 0.7] | 0.59 [0.5 to 0.8]
Statistical Analysis 1: Comparison: Patients Seen in the ED at Audit-and-feedback Sites vs Patients Seen in the ED at Control Sites; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Incident rate ratio = 0.88, 95% CI 2-sided [0.58 to 1.34]

5. Secondary Outcome: Percentage of Patient-visits Who Underwent Clostridium Difficile Testing More Than 24 Hours After But Within 30 Days of Their ED Visit
Description: Clostridium difficile testing is defined as a laboratory test for Clostridium difficile ordered more than 24 hours after but within 30-days of the patient's ED visit.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of visits tested
Arm/Group | Patients Seen in the ED at Audit-and-feedback Sites | Patients Seen in the ED at Control Sites
Number analyzed (Participants) | 51180 | 61912
percentage of visits tested
  Baseline: number analyzed (Participants) | 28016 | 33077
  Baseline | 0.60 [0.5 to 1.2] | 0.86 [0.7 to 1.2]
  Intervention period: number analyzed (Participants) | 23164 | 28835
  Intervention period | 0.69 [0.5 to 0.7] | 0.89 [0.7 to 1.2]
Statistical Analysis 1: Comparison: Patients Seen in the ED at Audit-and-feedback Sites vs Patients Seen in the ED at Control Sites; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Incident rate ratio = 0.83, 95% CI 2-sided [0.53 to 1.29]

6. Secondary Outcome: Percentage of Patient-visits Who Received Guideline Concordant Antimicrobial Management
Description: This outcome was assessed using blinded manual chart reviews in a randomly selected sample of patients that met inclusion criteria, as outlined in our study protocol. For this reason, the denominators for this outcome will not match the patient counts for the other outcomes. If a patient received an antimicrobial when indicated or did not receive an antimicrobial when not indicated, the patient was deemed to have received guideline-concordant management. During the baseline period, 497 charts were randomly selected for review, and 480 ultimately underwent adjudication. During the intervention period, 576 charts were randomly selected for review, and 455 underwent adjudication.
Time Frame: For the baseline and intervention periods, this outcome will be reported as the percentage of patients who received guideline-concordant management among the sample of qualifying ED visits that were randomly selected for manual chart review.
Population: For the Outcome Measure Data Table shown below, patient-visits were stratified by period (i.e. baseline and intervention period), and outcomes were compared across these two periods at intervention and control sites. Please see our statistical analysis plan for further details. For the intervention and control sites, the "overall number of participants analyzed" in the Arms/Groups table equals the sum of the "number analyzed" for the baseline and intervention periods, as shown below.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Seen in the ED at Audit-and-feedback Sites | Patients Seen in the ED at Control Sites
Number analyzed (Participants) | 470 | 465
Participants
  Baseline: number analyzed (Participants) | 240 | 240
  Baseline | 125 | 123
  Intervention: number analyzed (Participants) | 230 | 225
  Intervention | 166 | 131
Statistical Analysis 1: Comparison: Patients Seen in the ED at Audit-and-feedback Sites; Test type: Superiority; p = 0.001, Chi-squared
Statistical Analysis 2: Comparison: Patients Seen in the ED at Control Sites; Test type: Superiority; p = 0.13, Chi-squared

7. Secondary Outcome: Percentage of Patient-visits Prescribed an Antibiotic at Their ED Visit
Description: This outcomes is defined as the total number of antibacterial-prescribing visits divided by the total number of patient-visits. This metric will be calculated on a monthly basis for each site (2 intervention, 2 control). It will be calculated during the baseline and intervention periods. Therefore, each site will contribute 24 data points.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: % of visits prescribed an antibiotic
Arm/Group | Patients Seen in the ED at Audit-and-feedback Sites | Patients Seen in the ED at Control Sites
Number analyzed (Participants) | 51180 | 61912
% of visits prescribed an antibiotic
  Baseline | 20.8 [19.6 to 21.8] | 20.6 [18.7 to 22.2]
  Intervention | 18.2 [16.8 to 19.6] | 20.6 [19.4 to 21.9]
Statistical Analysis 1: Comparison: Patients Seen in the ED at Audit-and-feedback Sites vs Patients Seen in the ED at Control Sites; Test type: Superiority; p = 0.46, Regression, Logistic; Segmented regression analysis was conducted using generalized linear models to estimate change in monthly antibiotic prescription rates

ADVERSE EVENTS:
Time Frame: Outcomes were tracked for 30 days after each ED patient visit.
Description: Other adverse events consisted of Clostridioides difficile infections
Groups:
- Patients Seen at Audit-and-feedback ED Sites During Intervention Period: All patients seen in the EDs undergoing the audit-and-feedback intervention will be considered to have been exposed to the intervention. For this adverse event reporting section, we are reporting ED patient-visits during the intervention period at intervention sites.
  Because this study was not randomized, a more accurate assessment of adverse events would require a difference-in-differences analysis across the baseline and intervention periods while controlling for baseline differences between intervention and control sites. Such an analysis is described in our statistical analysis plan and will be reported in our published paper.
- Patients Seen at Control ED Sites During the Intervention Period: All patients seen in the EDs designated as control sites will be considered to have been part of the control group. For this adverse event reporting section, we are reporting ED patient-visits during the intervention period at control sites.
  Because this study was not randomized, a more accurate assessment of adverse events would require a difference-in-differences analysis across the baseline and intervention periods while controlling for baseline differences between intervention and control sites. Such an analysis is described in our statistical analysis plan and will be reported in our published paper.
- Patients Seen at Audit-and-feedback ED Sites During the Baseline Period: For this adverse event reporting section, we are only reporting ED patient-visits at intervention sites during the baseline period.
- Patients Seen at Control EDs During the Baseline Period: For this adverse event reporting section, we are reporting ED patient-visits at control sites during the baseline period.
Arm/Group | Patients Seen at Audit-and-feedback ED Sites During Intervention Period | Patients Seen at Control ED Sites During the Intervention Period | Patients Seen at Audit-and-feedback ED Sites During the Baseline Period | Patients Seen at Control EDs During the Baseline Period
All-Cause Mortality (participants affected / at risk) | 141/23164 | 176/28835 | 146/28016 | 197/33077
Serious Adverse Events (participants affected / at risk) | 1593/23164 | 1863/28835 | 1810/28016 | 2031/33077
Other Adverse Events (participants affected / at risk) | 11/23164 | 27/28835 | 193/28016 | 321/33077
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Seen at Audit-and-feedback ED Sites During Intervention Period (N=23164) | Patients Seen at Control ED Sites During the Intervention Period (N=28835) | Patients Seen at Audit-and-feedback ED Sites During the Baseline Period (N=28016) | Patients Seen at Control EDs During the Baseline Period (N=33077)
Hospitalization >24 hours after but within 30 days of ED visit (General disorders) | 1452 (1452) | 1687 (1687) | 1664 (1664) | 1834 (1834) — Any patient hospitalized more than 24 hours after but within 30 days of ED visit.
Mortality > 24 hours after ED visit and within 30 days of visit (General disorders) | 141 (141) | 176 (176) | 146 (146) | 197 (197)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Seen at Audit-and-feedback ED Sites During Intervention Period (N=23164) | Patients Seen at Control ED Sites During the Intervention Period (N=28835) | Patients Seen at Audit-and-feedback ED Sites During the Baseline Period (N=28016) | Patients Seen at Control EDs During the Baseline Period (N=33077)
Clostridioides difficile infection (Gastrointestinal disorders) | 11 (11) | 27 (27) | 193 (28016) | 321 (33077) — This reflects patients who were diagnosed and treated for an infection with Clostridioides difficile.

LIMITATIONS AND CAVEATS:
Because the study was not randomized, we cannot exclude temporal confounding or selection bias. By conducting a time-series analysis, we tried to account for confounders that may change over time, and by including a matched-control group, we tried to minimize the possibility of regression to the mean. Second, we cannot exclude the possibility that sites had any other processes in place that could have influenced our outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-24): https://cdn.clinicaltrials.gov/large-docs/67/NCT03349567/Prot_SAP_000.pdf